CLINICAL TRIAL: NCT01867112
Title: Physical Activity for Improving Quality of Life and Reducing Frailty in Advanced Age: Individually Tailored Program vs the General Guidelines Recommended by Offical Health Organizations.
Brief Title: Physical Activity for Improving Quality of Life and Reducing Frailty in Advanced Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYMC-26-13
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized Program (Active Comparator): Based on personal fitness an individualized physical activity program will be built and followed by each individual in the arm
  Interventions: Behavioral: Physical Activity
- General Physical Activity Guidelines (Active Comparator): The entire group of individuals in this arm will follow a physical activity program according to the General Physical Activity Guidelines
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Physical activity either by individualized program or general guidelines

SUMMARY:
Individuals of advanced age undergo both physical and cognitive deterioration. The aim of this study is to explore the connection between level of physical activity and health parameters, quality of life, and frailty.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65
* Able to undergo graded stress exam

Exclusion Criteria:

* All others

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Aerobic Fitness | One year
  Aerobic fitness will be measured with a graded stress exam

CONTACTS AND LOCATIONS:
Locations (1):
- Zinman College for Physical Education and Sport Sciences, Ramot Naftali, Israel